CLINICAL TRIAL: NCT07358039
Title: Impact of a Recruitment Maneuver After Closed Endotracheal Suctioning on End-expiratory Lung Volume in Mechanically Ventilated ICU Patients Assessed by Electrical Impedance Tomography
Brief Title: Effect of Post-suction Recruitment on Lung Volume in Mechanically Ventilated ICU Patients
Acronym: RESPIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-CHITS-013; 2025-A01845-44 (Other: ANSM)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mechanical Ventilation
Keywords: Endotracheal suction; Alveolar recruitment; Electrical impedance tomography; End-expiratory lung volume; Intensive care; Mechanical ventilation
MeSH Terms: interventions — Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Patients undergo closed-circuit endotracheal suctioning without a recruitment maneuver.
  Interventions: Procedure: Closed-circuit endotracheal suctioning
- B (Experimental): Patients undergo closed-circuit endotracheal suctioning immediately followed by a recruitment maneuver.
  Interventions: Procedure: Suction + Recruitment maneuver

INTERVENTIONS:
Procedure: Suction + Recruitment maneuver — After suctioning, a recruitment maneuver is applied consisting of an airway pressure of 30 cmH₂O maintained for 30 seconds, without changing the positive end-expiratory pressure.
  Arms: B
Procedure: Closed-circuit endotracheal suctioning — Standard closed-circuit endotracheal suctioning performed for less than 15 seconds without disconnecting the ventilator.
  Arms: A

SUMMARY:
Patients who are intubated and mechanically ventilated in the intensive care unit (ICU) require repeated endotracheal suctioning to remove airway secretions. Although this procedure is necessary, it can cause a temporary collapse of lung units (alveolar derecruitment), leading to a decrease in lung volume and impaired oxygenation.

A recruitment maneuver consists of briefly applying a higher airway pressure after suctioning in order to reopen collapsed lung areas and restore lung volume. However, the clinical benefit of performing a recruitment maneuver systematically after suctioning remains uncertain.

This study aims to evaluate whether performing a recruitment maneuver immediately after closed-circuit endotracheal suctioning improves lung volume compared with suctioning alone. Lung volume will be assessed using electrical impedance tomography (EIT), a non-invasive bedside imaging technique that allows real-time monitoring of lung aeration.

In a randomized crossover design, each patient will undergo two suctioning procedures: one followed by a recruitment maneuver and one without, in a random order. The main outcome will be the change in end-expiratory lung volume 15 minutes after suctioning. The results may help optimize ventilatory care in mechanically ventilated ICU patients.

DETAILED DESCRIPTION:
Endotracheal suctioning in mechanically ventilated ICU patients is a common procedure but is associated with alveolar derecruitment, resulting in a decrease in end-expiratory lung volume (EELV), deterioration of oxygenation, and potential lung injury.

A recruitment maneuver applied immediately after suctioning may reopen collapsed alveoli and restore lung volume, provided that sufficient positive end-expiratory pressure is maintained. However, available data are limited and conflicting, especially in adult ICU patients.

This prospective, randomized, open-label, single-center crossover trial will evaluate the physiological impact of a recruitment maneuver performed after closed-circuit endotracheal suctioning.

Each patient will receive two interventions in random order:

* Treatment A: closed-circuit endotracheal suctioning alone
* Treatment B: closed-circuit endotracheal suctioning followed immediately by a recruitment maneuver (airway pressure 30 cmH₂O for 30 seconds, with unchanged PEEP) Patients will be randomized to one of two sequences (AB or BA), with a 15-minute washout period between interventions.

Electrical impedance tomography (PulmoVista® V500) will be used to measure end-expiratory lung impedance, which reflects EELV. Functional residual capacity will be measured using nitrogen washout on a CARESCAPE R860 ventilator. Lung compliance and PaO₂/FiO₂ ratio will also be recorded.

Measurements will be obtained before suctioning and 15 minutes after each intervention. The primary endpoint is the percentage change in EELV at 15 minutes after suctioning between the two conditions.

A total of 32 mechanically ventilated ICU patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Covered by national health insurance
* Admitted to the intensive care unit
* Intubated and mechanically ventilated
* Neuromuscular blockade at inclusion
* Written informed consent obtained from a legally authorized representative or next of kin

Exclusion Criteria:

* Contraindication to electrical impedance tomography (e.g. pacemaker, implantable cardioverter-defibrillator, or implanted electrical stimulation device)
* Contraindication to recruitment maneuvers (e.g. emphysema, undrained pneumothorax, hemodynamic instability)
* Refractory intracranial hypertension
* Acute respiratory distress syndrome requiring prone positioning
* Pregnant or breastfeeding women
* Patients deprived of liberty or under legal protection
* Any condition judged by the investigator to interfere with study evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage change in end-expiratory lung volume (EELV) after suctioning | 15 minutes after endotracheal suctioning
  EELV assessed by end-expiratory lung impedance measured with electrical impedance tomography (PulmoVista® V500).

SECONDARY OUTCOMES:
Change in lung compliance | Baseline and 15 minutes after suctioning
  Measured from ventilator-derived respiratory mechanics.
Change in functional residual capacity (FRC) | Baseline and 15 minutes after suctioning
  Measured by nitrogen washout using the CARESCAPE R860 ventilator.
Change in PaO₂/FiO₂ ratio | Baseline and 15 minutes after suctioning
  Calculated from arterial blood gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril PERNOD, MD, Principal Investigator — Hôpital National d'Instruction des Armées (HNIA) Sainte-Anne, Toulon
Locations (1):
- Hôpital National d'Instruction des Armées Sainte-Anne, Toulon, VAR, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morrow B, Futter M, Argent A. A recruitment manoeuvre performed after endotracheal suction does not increase dynamic compliance in ventilated paediatric patients: a randomised controlled trial. Aust J Physiother. 2007;53(3):163-9. doi: 10.1016/s0004-9514(07)70023-5. PMID 17725473
- [Background] Kasim I, Gulyas M, Almgren B, Hogman M. A recruitment breath manoeuvre directly after endotracheal suction improves lung function: an experimental study in pigs. Ups J Med Sci. 2009;114(3):129-35. doi: 10.1080/03009730903177357. PMID 19736601
- [Background] Jesus AC, Figueiredo AM, Cordeiro ALL. Recruitment maneuvers in patients with acute respiratory distress syndrome: a systematic review and metanalysis. Einstein (Sao Paulo). 2024 Dec 16;22:eRW0372. doi: 10.31744/einstein_journal/2024RW0372. eCollection 2024. PMID 39699411
- [Background] Blakeman TC, Scott JB, Yoder MA, Capellari E, Strickland SL. AARC Clinical Practice Guidelines: Artificial Airway Suctioning. Respir Care. 2022 Feb;67(2):258-271. doi: 10.4187/respcare.09548. PMID 35078900